CLINICAL TRIAL: NCT05515068
Title: Registry For Children, Adolescents And Adults With Osteosarcoma And Biologically Related Bone Sarcomas (COSS-Registry)
Brief Title: Registry For Children, Adolescents And Adults With Osteosarcoma And Biologically Related Bone Sarcomas
Acronym: COSS-Registry
Status: Not yet recruiting | Type: Observational
Sponsor: Klinikum Stuttgart (Other)
Collaborators: Klinikum Kassel GmbH (COSS-Biobank) (Unknown)
Responsible Party: Sponsor
Other Study IDs: V.1.3 14.03.2022
Record Dates: First submitted 2022-08-16; First posted 2022-08-25 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Osteosarcoma; Bone Tumor; Bone Sarcoma; High Grade Sarcoma; Osteoblastic Osteosarcoma; Chondroblastic Osteosarcoma; Fibroblastic Osteosarcoma; Conventional Osteosarcoma; Conventional Central Osteosarcoma of Bone; Low Grade Central Osteosarcoma; Osseous Sarcoma; Osseous Tumor; Small Cell Osteosarcoma; Telangiectatic Osteosarcoma; Undifferentiated Pleomorphic Sarcoma; Parosteal Osteosarcoma; Periosteal Osteosarcoma; Extraskeletal Osteosarcoma; Recurrent Osteosarcoma; High Grade Surface Osteosarcoma; Osseous Angiosarcoma; Osseous Fibrosarcoma; Osseous Leiomyosarcoma; Osseous Dedifferentiated Chondrosarcoma; Osseous Mesenchymal Chondrosarcoma; Clear Cell Osteosarcoma
MeSH Terms: conditions — Osteosarcoma; Bone Neoplasms; Histiocytoma, Malignant Fibrous; Osteosarcoma, Juxtacortical

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — Tumor tissue and blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The Registry For Children, Adolescents And Adults With Osteosarcoma And Biologically Related Bone Sarcomas (COSS-Registry) is a non-interventional, multicentric, international, clinical and epidemiologic patient registry. The COSS-Registry collects key data on osteosarcomas or biologically related bone sarcomas. With that data collection we want to gain new scientific insights and results about this tumor disease, prognosis, surveillance and long-term effects.

Besides the data collection we would also like to foster the collection of biomaterial (tumor specimen and blood samples) for scientific research.

The stored material will be used to perform cell and molecular biological analyses to identify the causes of osteosarcoma, the prognosis and possible new treatment options.

As a starting point the donated biomaterial of registered patients will be analyzed firstly for the presence of a tumor predisposition by germline mutations.

In case of detected genetic variations that are related to the tumor disease and which may affect the patient's health and follow-up care (because of the potentially increased risk of developing other malignant tumors), affected patients will be informed and referred to genetic counseling.

Registry patients will be asked at the time of diagnosis if they wish to be informed about germline variants detected as part of the study procedures.

DETAILED DESCRIPTION:
Osteosarcomas are rare and malignant bone tumors with an incidence of only 200-300 diagnoses in Germany each year. The biological behaviour of the tumor is not well understood yet. Treatment options and survival prognosis have not improved for the last decades.

The planned collection of treatment and follow-up data of affected patients at the COSS-Registry has the goal to gain further insights about this tumor, to improve survival rates and to identify possible germline variants in tumor predisposition genes in any patient diagnosed with OS.

It is also necessary to foster research on the genetic and molecular biological characteristics of osteosarcoma by analyzing biomaterial samples (especially tumor tissue) for example to identify new therapy targets or to evaluate the response to and the adverse effects of chemotherapy with respect to the germline alterations.

Therefore a substantial amount of biomaterial has to be gathered and stored in a biobank. Accompanying to the COSS-Registry's data collection, biological samples taken from registered patients during routine measures and which are no longer required for further treatment will be stored in the COSS-Biobank.

The biological samples collected will be used to carry out genetic tests to check for an underlying tumor predisposition by germline mutations and for a next-generation sequencing of the whole genome. The goal of this project is to prospectively characterize the germline genetics in OS patients, to increase the understanding of the impact of germline alterations on the age of manifestation of OS, to evaluate the response to and the adverse effects of chemotherapy with respect to the germline alterations and to integrate germline investigation and counselling into the routine workup of any child, adolescent or young adult diagnosed with OS registered at the COSS-Registry.

In this way, affected patients will benefit from their participation in the COSS-Registry and COSS-Biobank.

ELIGIBILITY:
Inclusion Criteria:

* high-grade osteosarcoma (conventional and non-conventional)
* parosteal, periosteal or extraosseous osteosarcoma
* low grade central osteosarcoma
* (osseous) Undifferentiated pleomorphic sarcoma (UPS)
* (osseous) leiomyosarcoma
* (osseous) dedifferentiated chondrosarcoma
* (osseous) mesenchymal chondrosarcoma
* (osseous) fibrosarcoma
* (osseous) angiosarcoma
* informed consent

Exclusion Criteria:

* no informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients irrespective of gender, age and tumour location
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2032-03 (Estimated); Study Completion 2032-03 (Estimated)

PRIMARY OUTCOMES:
Data Collection | 20 years (There will be continous subgroup analyses through study completion.)
  Aims of the registry are the collection of clinical data to gain further insights about diagnosis, treatment, prognosis and risk factors of osteosarcoma and biologically related bone tumors.

SECONDARY OUTCOMES:
Reference Diagnostics | 20 years (Recruitment period)
  Aim of the registry is to give the frame for reference diagnostics.
Collection of biologic samples. | 20 years (Recruitment period)
  Aim of the registry is the collection of biomaterial.